CLINICAL TRIAL: NCT02880436
Title: Association of Air Quality and Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 28-292ex15/16
Record Dates: First submitted 2016-08-16; First posted 2016-08-26 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Air Pollution

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: air pollution — impact of various pollution agents above threshold and their correlation with acute myocardial infarctions are analyzed

SUMMARY:
Besides classical cardiovascular risk factors such as smoking, obesity, elevated cholesterol levels and diabetes there are also acute factors potentially triggering acute coronary events. The impact of various substances and air pollution are described.

Particulate matter, especially with small particle size (<2.5µm) has been shown to have a positive correlation with myocardial infarctions. However, other studies failed to show this correlation.

With respect to nitric oxydes the majority of published studies detected a significant correlation with myocardial infarction, too, although a highly ranked publication failed to show the same result. In addition data on the impact of sulfur dioxide and carbon monoxide concentration on cardiac events is very heterogeneous.

Published data indicates additive effects of age and other epidemiological variables suggesting the need of a multivariate analysis.

The rationale of the study is to test if the above mentioned air pollution factors have a significant and independent impact on the incidence of myocardial infarctions

DETAILED DESCRIPTION:
The analysis will be performed in a well characterized patient cohort of 12.000 myocardial infarctions within 10 years being invasively diagnosed at the catheterisation centers of the styrian capital Graz.

ELIGIBILITY:
Inclusion Criteria:

* myocardial infarction being confirmed or treated in the cathlab

Exclusion Criteria:

* none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with myocardial infarction being transfered to a cath lab either at the medical university of Graz or the department of cardiology at the state hospital Graz West
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2007-01; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
myocardial infarction | 1 day
  the number of myocardial infarctions of every day analysed in this study will be correlated with the respective values of air polluting substances

CONTACTS AND LOCATIONS:
Overall Officials: Dirk von Lewinski, MD, Principal Investigator — Dirk von Lewinski
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bhaskaran K, Hajat S, Haines A, Herrett E, Wilkinson P, Smeeth L. Effects of air pollution on the incidence of myocardial infarction. Heart. 2009 Nov;95(21):1746-59. doi: 10.1136/hrt.2009.175018. Epub 2009 Jul 26. PMID 19635723
- [Background] Sen T, Astarcioglu MA, Asarcikli LD, Kilit C, Kafes H, Parspur A, Yaymaci M, Pinar M, Tufekcioglu O, Amasyali B. The effects of air pollution and weather conditions on the incidence of acute myocardial infarction. Am J Emerg Med. 2016 Mar;34(3):449-54. doi: 10.1016/j.ajem.2015.11.068. Epub 2015 Dec 4. PMID 26742457
- [Background] Ruidavets JB, Cournot M, Cassadou S, Giroux M, Meybeck M, Ferrieres J. Ozone air pollution is associated with acute myocardial infarction. Circulation. 2005 Feb 8;111(5):563-9. doi: 10.1161/01.CIR.0000154546.32135.6E. PMID 15699276
- [Background] Barnett AG, Williams GM, Schwartz J, Best TL, Neller AH, Petroeschevsky AL, Simpson RW. The effects of air pollution on hospitalizations for cardiovascular disease in elderly people in Australian and New Zealand cities. Environ Health Perspect. 2006 Jul;114(7):1018-23. doi: 10.1289/ehp.8674. PMID 16835053